CLINICAL TRIAL: NCT03537235
Title: Randomized, Double-blind, Placebo-controlled Group, Single Center Study to Evaluate the Effect of 3 Months Policaptil Gel Retard Use on Postprandial Incretin Hormones Release and Satiety in Obese Women Regardless of Macronutrients Intake as Well as Body Mass Changes.
Brief Title: Evaluation of Libramed in Obesity Treatment
Acronym: ELOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELOT-14-2
Record Dates: First submitted 2018-02-09; First posted 2018-05-25 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Overweight and Obesity
Keywords: Libramed; Policaptil Gel retard; Overweigth; Obesity; Medical Device; glycemic profile; incretin
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Libramed (Experimental): 3 tablets of Libramed 2 twice a day 15 minutes before meals for 3 months.
  Interventions: Device: Libramed
- Placebo (Placebo Comparator): 3 tablets of Placebo 2 twice a day 15 minutes before meals for 3 months.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Libramed
  Other Names: Policaptil gel retard
  Arms: Libramed
Device: Placebo
  Other Names: Placebo-comparator
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled study aimed at evaluating the effects of a 3-months treatment with Policaptil Gel Retard on postprandial incretin hormones release and satiety in obese women

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled, parallel-group study.

This study will in made of 3 phases:

* The assessment of standard dose (3 tablets) of Libramed or placebo on the incretin hormones release and satiety sensation in obese women after ingestion of four test meal administered with one day interval - run-in period, to assess incretin hormones release and satiety sensation in obese women
* A double-blind phase in which the treament with Libramed/Placebo will be administered for 3 months.
* A post (3-months) treatment assessment of the incretin hormones release and satiety sensation after ingestion of four test meals - follow-up period.

During the screening visit (V1, Week -1) patients will be evaluated with regard to the inclusion and exclusion criteria that will permit their entry into the run-in period. The results of the laboratory analyses such as lipids, glucose and insulin levels needed to check subjects' eligibility at the time of randomization [baseline visit (V2)] will be performed at the screening visit. The run-in period starts on day 2 of the menstrual cycle and ends not later than 12 days of menstrual cycle.

During the four visits of run-in period (V2, V3, V4 and V5) will be assessed the effect of double-blind single dose of Libramed or placebo on postprandial incretin axis activity, glucose and triglycerides levels, satiety feeling and subsequent food consumption in relation to macronutrients content in test meals intake. During the visit V2 patient will be trained on diary completion.

On the first visit of this period (V5) patient previously randomized on the first visit of the run-in period (V2) will receive the first kit of Libramed or placebo. Each patient will self-administer 3 tablets of Libramed or placebo 2 times per day 15 minutes before breakfast and lunch. The dose of Libramed or placebo will be stable during the treatment period.

During the visit V5 patient will be trained on the Libramed or placebo self-administration, patient's diary completion and on diet and physical activity recommendation.

The follow-up period includes four visits (from V9 to V12), in the week immediately after the last intake of Libramed or placebo. The first visit of the follow-up period (V9) will take place the day immediately after the last intake of Libramed or placebo. The visits 9 to 12 (V9, V10, V11, V12) will take place with one day interval from each other, during the week after the last dose of Libramed or placebo use. On these visits the test meals will be administered and postprandial incretin axis, glucose and triglycerides levels as well as satiety feeling will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30.0-39.9 kg/m2,
* serum fasting glucose and insulin in normal ranges (- glucose ≤ 100 mg/dl, insulin ≤ 15 uIU/ml)
* HOMA-IR < 2.5 (normal range for insulin sensitivity among Polish population),
* stable body mass in the last 3 months (not more than 2 kg),
* do not use any hypocaloric diet in the last 6 months,
* not changed then realized before physical activity in the last 3 months,
* the lack of any known comorbidities,
* do not use any drugs including contraceptive
* capability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* All chronic and acute disease of the digestive tract in medical history,
* smoking,
* more than 3 alcoholic drinks per week (bear, glass of wine, and 50 ml vodka)
* no patient co-operation.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of postprandial incretin axis activity | day 1 to day 91
  incretin axis activity
Evaluation of postprandial glycemic profile | day 1 to day 91
  blood samples for glucose measurements ( will be collected on visits 1, 2, 3, 4 and 8, 9, 10, 11, 12 on the fasting state and during the postprandial 6-hours observations (6 time collections 1, 2, 3, 4, 5, 6 hours after the test meal intake).
Evaluation of triglycerides levels | day 1 to day 91
  Blood samples for triglycerides measurements will be collected on visits 1, 2, 3, 4 and 8, 9,10,11,12 on the fasting state and during the postprandial 6-hours observations (6 time collections 1, 2, 3, 4, 5, 6 hours after the test meal intake).
Evaluation of satiety feeling | day 1 to day 91
  On visit 2 and 8 the subjective fasting satiety and hunger sensation will be assessed on the basis of visual analogue scale (VAS) at the baseline (V2) and at the end of the double-blind treatment period (V8). In addition fasting and postprandial VAS scales will be filled by the test 5 minutes before Libramed product or placebo administration, 5 minutes before eating a test meal and 1, 2, 3, 4, 5, 6 hour after test meal consumption during the run-in period (V5) and follow-up period (V9-V12).

SECONDARY OUTCOMES:
Evaluation of postprandial incretin axis activity - single dose assessment | day -6 to day 1
  incretin axis activity in postprandial 6-hours observations (6 time collections 1, 2, 3, 4, 5, 6 hours after the test meal intake).
Evaluation of postprandial glycemic profile - single dose assessment | day -6 to day 1
  Blood samples for glucose measurements will be collected on visits 1, 2, 3, 4 and during the postprandial 6-hours observations (6 time collections 1, 2, 3, 4, 5, 6 hours after the test meal intake).
Evaluation of postprandial triglycerides - single dose assessment | day -6 to day 1
  Blood samples for triglycerides measurements will be collected on visits 1, 2, 3, 4 and during the postprandial 6-hours observations (6 time collections 1, 2, 3, 4, 5, 6 hours after the test meal intake).
Evaluation of satiety feeling - single dose assessment | day -6 to day 1
  Fasting and postprandial 100 mm Visual Analog Scale (VAS) (from "no symptoms" to "overwhelming symptoms") will be filled by the test 5 minutes before Libramed product or placebo administration, 5 minutes before eating a test meal and 1, 2, 3, 4, 5, 6 hour after test meal consumption during the run-in period (V5).
Evaluation of reduction in subsequent food consumption in relation to macronutrients content in test meals. | day -6 and day 84
  On visit 2 and 8 the food preferences will be assessed at the beginning and end of the study with its own survey takes into account the ten products of protein, fat and carbohydrate. To each product is assigned one point. Total points in the products group will be indicative for food preferences.
Body Mass assessment | day-7, day-6, day-4, day-2, day0, day28, day56, day84, day85, day87, day89, day91
  Body mass will be measured on each study visit.
Fat Mass assessment | day-7, day-6, day-4, day-2, day0, day28, day56, day84, day85, day87, day89, day91
  Fat mass will be measured on each study visit.
Waist circumference assessment | day-7, day-6, day-4, day-2, day0, day28, day56, day84, day85, day87, day89, day91
  waist circumference will be measured on each study visit.
Fasting glucose levels assessment | day 84 to day 91
  glucose measurements will be collected on visits 8, 9, 10, 11, 12 on the fasting state.
Fasting insulin levels assessment | day 84 to day 91
  insulin measurements will be collected on visits 8, 9, 10, 11, 12 on the fasting state.
Fasting lipids levels assessment | day 84 to day 91
  lipids measurements will be collected on visits 8, 9, 10, 11, 12 on the fasting state.
Fasting incretin axis activity | day 84 to day 91
  incretin axis activity measurements will be collected on visits 8, 9, 10, 11, 12 on the fasting state.
Safety and tolerability | day -7 to day 91
  Clinical safety will be assessed by physical examination at the V1, V4, V8, V12.

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolic Management Center "LINIA", Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.aboca.com/en/our-products/fitomagra-libramed